CLINICAL TRIAL: NCT01697787
Title: Efficacy of Amodiaquine-Artesunate (ASAQ) and Artemether-Lumefantrine (AL) for the Treatment of Uncomplicated Falciparum Malaria in Nanoro, Burkina Faso
Brief Title: Amodiaquine-Artesunate & Artemether-Lumefantrine Efficacy in Burkina Faso
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Muraz (Other)
Collaborators: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Principal Investigator, Tinto Halidou, PharmD, PhD, Centre Muraz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM/CRUN0012
Record Dates: First submitted 2012-09-29; First posted 2012-10-02 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Malaria
Keywords: Treatment, diagnosis
MeSH Terms: conditions — Malaria; Disease | interventions — amodiaquine, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Amodiaquine-Artesunate (Other): ASAQ is produced by Sanofi-Aventis as CoarsucamTM and as artesunate-amodiaquine Winthrop®
  Interventions: Drug: Amodiaquine-Artesunate
- Artemether-Lumefantrine (Other): AL (tablets containing 20 mg of artemether and 120 mg of lumefantrine) is produced by Novartis
  Interventions: Drug: Artemether-lumefantrine

INTERVENTIONS:
Drug: Amodiaquine-Artesunate — If necessary, the study drug will be crushed, dissolved in water and squirted into the mouth using a spoonful. Administration of the treatments will be directly observed. After drug administration, patients will be kept for at least 30 minutes in the clinic. A dose will be repeated in full if vomiting occurs within 30 minutes of administration and halved if vomiting is between 30 minutes and 1 hour post dosing.
  Other Names: ASAQ Winthrop, Coarsucam
  Arms: Amodiaquine-Artesunate
Drug: Artemether-lumefantrine — If necessary, the study drug will be crushed, dissolved in water and squirted into the mouth using a spoonful. Administration of the treatments will be directly observed. After drug administration, patients will be kept for at least 30 minutes in the clinic. A dose will be repeated in full if vomiting occurs within 30 minutes of administration and halved if vomiting is between 30 minutes and 1 hour post dosing.
  Other Names: Coartem, Riamet
  Arms: Artemether-Lumefantrine

SUMMARY:
This is a two-arm study aiming at recruiting 150 patients to assess the efficacy of Amodiaquine-Artesunate (ASAQ) and Artemether-Lumefantrine (AL) in patients with a microscopy positive diagnosis of malaria in Nanoro, Burkina Faso and assess the performance of the Rapid Diagnosis Tests (RDTs) compared to the microscopy.

DETAILED DESCRIPTION:
Study background and purpose

* Resistance to usual drugs was widespread and has required a change of the malaria treatment by several countries
* Several countries have changed their first-line treatments to ACTs; mainly AL and ASAQ. & have adopted the use of RDTs prior to treatment
* Indeed, this contributes to decrease the number of unnecessary treatments and thus improve the management of malaria cases.
* In February 2005, Burkina Faso changed its national drug policy from Chloroquine to Amodiaquine-Artesunate (ASAQ) and Artemether-Lumefantrine (AL)
* the country has also implemented the strategy of using the Rapid Diagnosis Tests (RDTs) for the diagnosis of malaria prior to treatment
* Though endemic countries are being encouraged to implement RDTs, choosing a particular RDT is not easy as several brands are available on the market.
* In addition, little information on the performance of RDTs in Africa is available and recently quality problems have been reported with some RDTs.
* In this context, it is important to locally assess the performance of RDTs compared with the microscopy, which is the gold standard for the malaria diagnosis and to assess the efficacy of the new drugs used for malaria treatment

This is a phase IV two-arm randomized open-label study aiming at recruiting 150 patients to assess the efficacy of ASAQ and AL in patients with a microscopy positive diagnosis of malaria in Nanoro, Burkina Faso and assess the performance of the RDT compared to the microscopy

ELIGIBILITY:
Inclusion Criteria:

* Age above 6 months,
* eight above 5 kg;
* Positive blood slide (parasitaemia ≥ 2,000/μL to 200,000/μL) with Plasmodium falciparum monospecific infection ;
* Fever (axillary temperature above 37.5 °C) or history of fever in the preceding 24 hours;
* Haemoglobin value above or equal 5.0 g/dL
* Signed informed consent;
* Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

* Participation in any other investigational drug study (antimalarial or others) during the previous 30 days
* Known hypersensitivity to the study drugs
* Severe malaria
* Danger signs: not able to drink or breast-feed, vomiting (> twice in 24hours), recent history of convulsions (more than 1 in 24h), unconscious state, unable to sit or stand;
* Known intercurrent illness or any condition (cardiac, renal, hepatic diseases) which would place the subject at undue risk or interfere with the results of the study.
* Severe malnutrition (defined as weight for height less than 70% of the median NCHS/WHO reference)
* Known pregnancy

Ages: 6 Months to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Rate of treatment failures | 28 days
  The rate of the two ACTs treatment failures at day 28: all treatment failures, both parasitological and clinical (positive blood slide at day 28)

SECONDARY OUTCOMES:
RDT performance Vs microscopy | 28 days
  The proportion of discrepancies between the RDT and the microscopy results

OTHER OUTCOMES:
Fever clearance time (FCT) Fever Clearance Time | 28 days
  Fever clearance time will be defined as the time (in days) from the time of the drug administration to the first two consecutive measurements on 2 different days of axillary temperature below 37.5°C
Gametocytes carriage | 28 days
  Gametocytes carriage including the estimation of the prevalence and density

CONTACTS AND LOCATIONS:
Overall Officials: Halidou Tinto, PharmD, PhD, Study Director — IRSS/Centre Muraz
Locations (1):
- Clinical Reaserch Unit, Nanoro, Boulkiemdé, Burkina Faso